CLINICAL TRIAL: NCT05537025
Title: A Phase 1/2a Study Evaluating the Effects of ARO-MMP7 Inhalation Solution in Healthy Subjects and Patients With Idiopathic Pulmonary Fibrosis
Brief Title: Study of ARO-MMP7 Inhalation Solution in Healthy Subjects and Patients With Idiopathic Pulmonary Fibrosis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Arrowhead Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AROMMP7-1001; 2023-504964-41 (EudraCT Number)
Record Dates: First submitted 2022-09-08; First posted 2022-09-13 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- ARO-MMP7 (Experimental): single or multiple doses of ARO-MMP7 by inhalation of nebulized solution
  Interventions: Drug: ARO-MMP7 Inhalation Solution
- Placebo (Placebo Comparator): single or multiple doses of placebo by inhalation of nebulized solution
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ARO-MMP7 Inhalation Solution — ARO-MMP7 by inhalation of nebulized solution
  Arms: ARO-MMP7
Drug: Placebo — Calculated volume of normal saline (0.9% NaCl) to match active treatment by inhalation of nebulized solution
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, pharmacokinetics (PK) and pharmacodynamics (PD) of ARO-MMP7 in normal healthy volunteers (NHVs) and in participants with idiopathic pulmonary fibrosis (IPF). The study will initiate with NHVs receiving single ascending doses of ARO-MMP7. Following evaluation of safety and pharmacodynamic (PD) data, participants will receive multiple doses of ARO-MMP7.

ELIGIBILITY:
Inclusion Criteria (NHVs):

* Normal pulmonary function tests at Screening
* Normal electrocardiogram (ECG) at Screening
* Non-smoking
* Female participants cannot be pregnant or lactating
* Male and female participants of childbearing potential must agree to use highly effective contraception and must not donate eggs/sperm during the study and for at least 90 days following end of study or last dose of study drug, whichever is later.

Inclusion Criteria (IPF Participants):

* Age ≥ 45 years at Screening
* Clinical diagnosis consistent with IPF based upon established criteria confirmed by review of high-resolution computed tomography (HRCT) and surgical lung biopsy findings (if available)
* Safely able to undergo bronchoscopy
* Stable IPF disease at Screening with minimum life expectancy of ≥ 12 months from Screening
* Female participants cannot be pregnant or lactating
* Male and female participants of childbearing potential must agree to use highly effective contraception and must not donate eggs/sperm during the study and for at least 90 days following end of study or last dose of study drug, whichever is later.

Exclusion Criteria (NHVs):

* Acute lower respiratory infection within 30 days prior to first dose or acute upper respiratory infection within 7 days prior to first dose
* Positive COVID-19 test during Screening window
* Any history of chronic pulmonary disease or anaphylaxis
* Human immunodeficiency virus (HIV) infection, seropositive for hepatitis B virus (HBV), seropositive for hepatitis C virus (HCV)
* Uncontrolled hypertension
* History of significant cardiac disease
* History of major surgery within 12 weeks prior to first dose
* Unwilling to limit alcohol consumption to within moderate limits for the duration of the study
* Use of illicit drugs
* Use of an investigational agent or device within 30 days prior to first dose

Exclusion Criteria (IPF Participants):

* Interstitial lung disease (ILD) associated with known primary cause
* Positive COVID-19 test during Screening window
* IPF exacerbation within 6 weeks prior to first dose
* Lower respiratory tract infection requiring antibiotics or antivirals within 30 days prior to first dose
* Smoking cigarettes or e-cigarettes within 3 months prior to first dose
* Use of systemic corticosteroid therapy within 30 days prior to first dose
* Initiation or cessation of antifibrotic therapy or change of antifibrotic dose regimen within 10 weeks prior to first dose
* Any history of lung transplant or plan to undergo transplant during the course of the study
* Any concomitant pulmonary disease that could interfere with the evaluation of the study drug or interpretation of patient safety or study results
* HIV infection, seropositive for HBV, seropositive for HCV
* Uncontrolled hypertension
* History of significant cardiac disease
* History of major surgery within 12 weeks prior to first dose
* Unwilling to limit alcohol consumption to within moderate limits for the duration of the study
* Use of illicit drugs
* Use of an investigational agent or device within 30 days prior to first dose

Note: additional inclusion/exclusion criteria may apply per protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2023-01-30 (Actual); Primary Completion 2025-09-05 (Actual); Study Completion 2025-09-05 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Treatment-Emergent Adverse Events (TEAEs) Over Time | From first dose of study drug through the end of study (EOS; up to 85 days, or until sputum MMP7 protein concentration is ≥ 70% of the baseline value, whichever is later)

SECONDARY OUTCOMES:
Change From Baseline Over Time in Forced Expiratory Volume (FEV1) | Baseline through EOS (up to 85 days, or until serum MMP7 protein concentration is ≥ 70% of the baseline value, whichever is later)
Change From Baseline Over Time in Forced Vital Capacity (FVC) | Baseline through EOS (up to 85 days, or until serum MMP7 protein concentration is ≥ 70% of the baseline value, whichever is later)
Change From Baseline Over Time in Diffusing Capacity for Carbon Monoxide (DLCO) | Baseline through EOS (up to 85 days, or until serum MMP7 protein concentration is ≥ 70% of the baseline value, whichever is later)
PK of ARO-MMP7: Maximum Observed Plasma Concentration (Cmax) | single dose phase: up to 168 hours post-dose; multiple dose phase: up to 6 hours post-dose on Days 1 and 15 or 29, 24 hours post-dose on Days 2 and 30, and (IPF only) Days 8, 22, and 36
PK of ARO-MMP7: Area Under the Plasma Concentration versus Time Curve from Zero to 24 Hours (AUC0-24) | single dose phase: up to 168 hours post-dose; multiple dose phase: up to 6 hours post-dose on Days 1 and 15 or 29, 24 hours post-dose on Days 2 and 30, and (IPF only) Days 8, 22, and 36
PK of ARO-MMP7: Area Under the Plasma Concentration versus Time Curve from Zero to the Last Quantifiable Plasma Concentration (AUClast) | single dose phase: up to 168 hours post-dose; multiple dose phase: up to 6 hours post-dose on Days 1 and 15 or 29, 24 hours post-dose on Days 2 and 30, and (IPF only) Days 8, 22, and 36
PK of ARO-MMP7: Area Under the Plasma Concentration versus Time Curve from Zero to Infinity (AUCinf) | single dose phase: up to 168 hours post-dose; multiple dose phase: up to 6 hours post-dose on Days 1 and 15 or 29, 24 hours post-dose on Days 2 and 30, and (IPF only) Days 8, 22, and 36
PK of ARO-MMP7: Terminal Elimination Half-Life (t1/2) | single dose phase: up to 168 hours post-dose; multiple dose phase: up to 6 hours post-dose on Days 1 and 15 or 29, 24 hours post-dose on Days 2 and 30, and (IPF only) Days 8, 22, and 36
PK of ARO-MMP7: Apparent Systemic Clearance (CL/F) | single dose phase: up to 168 hours post-dose; multiple dose phase: up to 6 hours post-dose on Days 1 and 15 or 29, 24 hours post-dose on Days 2 and 30, and (IPF only) Days 8, 22, and 36
PK of ARO-MMP7: Apparent Terminal Phase Volume of Distribution (VZ/F) | single dose phase: up to 168 hours post-dose; multiple dose phase: up to 6 hours post-dose on Days 1 and 15 or 29, 24 hours post-dose on Days 2 and 30, and (IPF only) Days 8, 22, and 36
PK of ARO-MMP7: Recovery of Unchanged Drug in Urine Over 0 to 24 Hours (Amount excreted; Ae) in NHVs | single dose phase: up to 168 hours post-dose; multiple dose phase: up to 6 hours post-dose on Days 1 and 15 or 29, 24 hours post-dose on Days 2 and 30
PK of ARO-MMP7: Percentage of Administered Drug Recovered in Urine Over 0 to 24 Hours in NHVs | single dose phase: up to 168 hours post-dose; multiple dose phase: up to 6 hours post-dose on Days 1 and 15 or 29, 24 hours post-dose on Days 2 and 30
PK of ARO-MMP7: Renal Clearance (CLr) in NHVs | single dose phase: up to 168 hours post-dose; multiple dose phase: up to 6 hours post-dose on Days 1 and 15 or 29, 24 hours post-dose on Days 2 and 30

CONTACTS AND LOCATIONS:
Locations (19):
- Denmark (2):
  - Research Site 1, Copenhagen
  - Research Site 2, Odense
- Italy (5):
  - Research Site 1, Ancona
  - Research Site 2, Florence
  - Research Site 3, Milan
  - Research Site 4, Milan
  - Research Site 5, Milan
- New Zealand (2):
  - Research Site 1, Auckland
  - Research Site 2, Christchurch
- South Korea (3):
  - Research Site 2, Seoul
  - Research Site 3, Soeul
  - Research Site 1, Ulsan
- Spain (3):
  - Research Site 3, Santander, Cantabria
  - Research Site 1, Barcelona
  - Research Site 2, Oviedo
- United Kingdom (4):
  - Research Site 1, Birmingham
  - Research Site 2, Edinburgh
  - Research Site 4, Manchester
  - Research Site 3, Manchester

IPD SHARING:
Plan to Share IPD: No